CLINICAL TRIAL: NCT03546816
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Pruritus in Adults With Prurigo Nodularis
Brief Title: Study of the Efficacy, Safety and Tolerability of Serlopitant for the Treatment of Pruritus (Itch) With Prurigo Nodularis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI-105
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pruritus; Prurigo Nodularis
MeSH Terms: conditions — Pruritus | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 mg Serlopitant Tablets (Experimental)
  Interventions: Drug: 5mg Serlopitant Tablets
- Matching Placebo Tablets (Placebo Comparator)
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: 5mg Serlopitant Tablets — Serlopitant Tablets
  Other Names: VPD-737
  Arms: 5 mg Serlopitant Tablets
Drug: Placebo Tablets — Placebo Tablets
  Arms: Matching Placebo Tablets

SUMMARY:
Study of the efficacy, safety, and tolerability of serlopitant for the treatment of pruritus in adults with prurigo nodularis

ELIGIBILITY:
Inclusion Criteria (Subjects must meet the following criteria to be randomized into the study:

1. Male or female, age 18 years or older at consent.
2. Prurigo nodularis (PN), with at least ten nodules on at least two different body surface areas.
3. Idiopathic PN, or an identified pruritic condition associated with the PN with persistent pruritus despite at least 6 weeks of optimized and stable treatment of the underlying condition.
4. The worst pruritus is identified as within the areas of the PN lesions, with a Worst-Itch Numeric Rating Scale (WI-NRS) score in the 24-hour period prior to the Screening visit, and average weekly WI-NRS score in each of the 2 weeks prior to Baseline visit indicating an appropriate pruritus level for the study.
5. Female subjects of childbearing potential must be willing to practice highly effective contraception until 5 weeks after last dose of study drug.
6. Willing and able to complete daily eDiary entries within a consistent timeframe for the duration of the study.
7. Willing and able to comply with study visits and study related requirements including providing written informed consent.

Exclusion Criteria (Subjects who meet any of the following criteria are not eligible for participation in the study):

1. Prior treatment with serlopitant.
2. Active pruritic skin disease, other than PN, within 6 months (with the exception of acute dermatoses such as contact dermatitis, sunburn, viral exanthem, which have been resolved for longer than 4 weeks).
3. Treatment with any of the following therapies within 4 weeks.

   1. Other neurokinin-1 receptor antagonists (e.g., aprepitant, fosaprepitant, rolapitant).
   2. Systemic or topical immunosuppressive/immunomodulatory therapies.
   3. Systemic therapies with recognized anti-pruritic properties.
   4. Strong cytochrome-P 3A4 inhibitors.
   5. Use of an indoor tanning facility, or natural sun exposure resulting in significant tanning or sunburn.
4. Treatment with topical anti-pruritic therapies within 2 weeks.
5. Treatment with biologic therapies within 8 weeks or 5 half-lives, whichever is longer.
6. Treatment with any investigational therapy within 4 weeks (8 weeks for investigational biologic therapies) or 5 half-lives, whichever is longer.
7. Serum creatinine, total bilirubin, alanine aminotransferase or aspartate aminotransferase > 2.5 times the upper limit of normal during screening.
8. Untreated or inadequately treated thyroid adrenal, or pituitary nodules or disease, or history of thyroid malignancy.
9. Malignancy within 5 years prior to enrollment (exception for non-melanoma cutaneous malignancies).
10. Relevant major psychiatric diagnosis in the past 3 years, such as major depressive disorder, bipolar disorder, schizophrenia, psychotic disorder, intellectual disability, severe alcohol use disorder.
11. Documented history of parasitic infection, including skin parasites such as scabies, within 8 weeks.
12. Any medical condition or disability that could interfere with the assessment of safety or efficacy in this study or compromise the safety of the subject.
13. History of hypersensitivity to serlopitant or any of its components.
14. Currently pregnant or breastfeeding or planning to become pregnant during the study.
15. Planned or anticipated major surgical procedure or other activity that would interfere with the subject's ability to comply with protocol-mandated assessments during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Study Site 504, Birmingham, Alabama
  - Study Site 533, Rogers, Arkansas
  - Study Site 204, Fremont, California
  - Study Site 383, North Hollywood, California
  - Study Site 356, San Diego, California
  - Study Site 514, Santa Ana, California
  - Study Site 501, Aventura, Florida
  - Study Site 210, Coral Gables, Florida
  - Study Site 534, Fort Lauderdale, Florida
  - Study Site 531, Miami, Florida
  - Study Site 530, Miami, Florida
  - Study Site 222, North Miami Beach, Florida
  - Study Site 510, Newnan, Georgia
  - Study Site 388, Skokie, Illinois
  - Study Site 228, Louisville, Kentucky
  - Study Site 527, New Orleans, Louisiana
  - Study Site 525, Glenn Dale, Maryland
  - Study Site 379, Boston, Massachusetts
  - Study Site 506, Ann Arbor, Michigan
  - Study Site 515, Detroit, Michigan
  - Study Site 371, Saint Joseph, Missouri
  - Study Site 528, St Louis, Missouri
  - Study Site 227, Omaha, Nebraska
  - Study Site 526, Henderson, Nevada
  - Study Site 201, East Windsor, New Jersey
  - Study Site 529, Verona, New Jersey
  - Study Site 507, Brooklyn, New York
  - Study Site 508, Buffalo, New York
  - Study Site 500, New York, New York
  - Study Site 517, New York, New York
  - Study Site 341, High Point, North Carolina
  - Study Site 516, Bexley, Ohio
  - Study Site 509, Cleveland, Ohio
  - Study Site 524, Dublin, Ohio
  - Study Site 112, Tulsa, Oklahoma
  - Study Site 523, Philadelphia, Pennsylvania
  - Study Site 522, Pittsburgh, Pennsylvania
  - Study Site 345, Johnston, Rhode Island
  - Study Site 511, Knoxville, Tennessee
  - Study Site 805, Nashville, Tennessee
  - Study Site 365, Austin, Texas
  - Study Site 520, Bellaire, Texas
  - Study Site 502, Dallas, Texas
  - Study Site 224, Houston, Texas
  - Study Site 359, Pflugerville, Texas
  - Study Site 361, San Antonio, Texas
  - Study Site 226, Webster, Texas
  - Study Site 806, Spokane, Washington
  - Study Site 532, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 sites in United States from 02 May 2018 to 14 February 2020. All subjects who met the study entry criteria were randomized in a 1:1 ratio to receive once-daily oral doses of serlopitant 5 mg or placebo for 10 weeks.
Pre-assignment Details: During the screening period (2-4 weeks), all subjects were evaluated for eligibility and assessed for conditions associated with chronic pruritus. Subjects were to complete an electronic diary (eDiary) during screening visit.
Groups:
- Serlopitant 5 mg: Randomized subjects received serlopitant 5 mg as an initial loading dose (3 tablets orally) on Day 1, the first day of the treatment period. Thereafter, starting on Day 2, subjects were instructed to take 1 tablet orally per day.
- Placebo: Randomized subjects received placebo as an initial loading dose (3 tablets orally) on Day 1, the first day of the treatment period. Thereafter, starting on Day 2, subjects were instructed to take 1 tablet orally per day.
Period: Overall Study
Arm/Group | Serlopitant 5 mg | Placebo
Started | 142 | 143
Completed | 121 | 124
Not Completed | 21 | 19
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 2 | 4
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 8 | 10
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serlopitant 5 mg | Placebo | Total
Number analyzed (Participants) | 142 | 143 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Three subjects were excluded in the serlopitant 5 mg arm and 2 subjects were excluded in the placebo arm due to no evidence of subject dosing and/or no post-Baseline assessment/treatment emergent adverse event (TEAE).
  Years
    number analyzed (Participants) | 139 | 141 | 280
    (all) | 58.7 (13.54) | 56.0 (12.99) | 57.4 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Three subjects were excluded in the serlopitant 5 mg arm and 2 subjects were excluded in the placebo arm due to no evidence of subject dosing and/or no post-Baseline assessment/TEAE.
  Participants
    number analyzed (Participants) | 139 | 141 | 280
    Female | 92 | 89 | 181
    Male | 47 | 52 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three subjects were excluded in the serlopitant 5 mg arm and 2 subjects were excluded in the placebo arm due to no evidence of subject dosing and/or no post-Baseline assessment/TEAE.
  Participants
    number analyzed (Participants) | 139 | 141 | 280
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 6 | 11 | 17
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 27 | 33 | 60
    White | 102 | 91 | 193
    More than one race | 3 | 5 | 8
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Worst-Itch Numeric Rating Scale 4-point Responder at Week 10
Description: During the study, Worst Itch Numeric Rating Scale (WI-NRS) assessments were reported by the subject via eDiary once daily from screening/mid-screening visit through the follow-up visit. The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subjects were asked to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores indicated greater itch intensity. Subjects were considered responders if they had at least a 4-point reduction from baseline in weekly average WI-NRS at Week 10.
Time Frame: At Week 10
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Number; unit: Percentage of subjects
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Percentage of subjects | 26.45 | 20.31
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; Test type: Superiority; p = 0.229, Cochran-Mantel-Haenszel — P-value from a Cochran-Mantel-Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation

2. Secondary Outcome: Percent of Subjects With WI-NRS 4-point Responder at Week 4
Description: During the study, WI-NRS assessments were reported by the subject via eDiary once daily from screening/mid-screening visit through the follow-up visit. The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subjects were asked to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores indicated greater itch intensity.
Time Frame: At Week 4
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Number; unit: Percentage of subjects
Groups:
- Serlopitant 5 mg: Randomized subjects received Serlopitant 5 mg as an initial loading dose (3 tablets orally) on Day 1, the first day of the treatment period. Thereafter, starting on Day 2, subjects were instructed to take 1 tablet orally per day on an outpatient basis.
- Placebo: Randomized subjects received placebo as an initial loading dose (3 tablets orally) on Day 1, the first day of the treatment period. Thereafter, starting on Day 2, subjects were instructed to take 1 tablet orally per day on an outpatient basis.
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Percentage of subjects | 17.66 | 7.80
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel — P-value from a CMH test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation

3. Secondary Outcome: Percent of Subjects With WI-NRS 4-point Responder at Week 2
Description: as for outcome 2
Time Frame: At Week 2
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Number; unit: Percentage of subjects
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Percentage of subjects | 8.45 | 4.93
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; Test type: Superiority; p = 0.236, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in WI-NRS at Weeks 2, 4, 6, and 10
Description: as for outcome 2
Time Frame: At Weeks 2, 4, 6, and 10
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Score on a scale
  Change from Baseline at Week 2 | -1.30 (1.725) | -0.96 (1.740)
  Change from Baseline at Week 4 | -1.82 (2.226) | -1.32 (2.248)
  Change from Baseline at Week 6 | -2.13 (2.436) | -1.65 (2.460)
  Change from Baseline at Week 10 | -2.47 (2.633) | -2.06 (2.612)
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; At Week 2; Test type: Superiority; p = 0.083, ANCOVA — P-values, least squares means (LS Mean) and standard deviations (LS SD) from an analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate
Statistical Analysis 2: Comparison: Serlopitant 5 mg vs Placebo; At Week 4; Test type: Superiority; p = 0.049, ANCOVA — P-values, LS mean and SD from ANCOVA with treatment group and stratification factor as fixed effects, and baseline value as a covariate
Statistical Analysis 3: Comparison: Serlopitant 5 mg vs Placebo; At Week 6; Test type: Superiority; p = 0.081, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Serlopitant 5 mg vs Placebo; At Week 10; Test type: Superiority; p = 0.157, ANCOVA — [p-value comment as in outcome 4, analysis 2]

5. Secondary Outcome: Percent of Subjects With WI-NRS 3-point Responder at Weeks 2, 4, and 10
Description: During the study, WI-NRS assessments were reported by the subject via eDiary once daily from screening/mid-screening visit through the follow-up visit. The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subjects were asked to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores indicated greater itch intensity. For the 3-point responder rate, subjects were considered responders if they had at least a 3-point reduction between baseline and the corresponding week.
Time Frame: At Weeks 2, 4, and 10
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Number; unit: Percentage of subjects
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Percentage of subjects
  Percentage of responders at Week 2 | 14.79 | 9.27
  Percentage of responders at Week 4 | 23.32 | 14.31
  Percentage of responders at Week 10 | 35.58 | 27.83
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; At Week 2; Test type: Superiority; p = 0.151, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Serlopitant 5 mg vs Placebo; At Week 4; Test type: Superiority; p = 0.052, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Serlopitant 5 mg vs Placebo; At Week 10; Test type: Superiority; p = 0.175, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline in Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A) to Weeks 2, 4, and 10
Description: The IGA PN-A is an instrument used to assess the overall activity of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 (clear) to 4 (severe). Higher scores indicate severe prurigo nodularis.
Time Frame: At Weeks 2, 4, and 10
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Score on a scale
  Change from Baseline at Week 2 | -0.3 (0.71) | -0.3 (0.71)
  Change from Baseline at Week 4 | -0.6 (0.81) | -0.4 (0.81)
  Change from Baseline at Week 10 | -0.7 (0.99) | -0.6 (0.99)
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; At Week 2; Test type: Superiority; p = 0.475, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 2: Comparison: Serlopitant 5 mg vs Placebo; At Week 4; Test type: Superiority; p = 0.020, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Serlopitant 5 mg vs Placebo; At Week 10; Test type: Superiority; p = 0.492, ANCOVA — [p-value comment as in outcome 4, analysis 2]

7. Secondary Outcome: Change From Baseline in Investigator's Global Assessment of PN Stage (IGA PN-S) to Weeks 2, 4, and 10
Description: The IGA PN-S is an instrument used to assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 (clear) to 4 (severe). Higher scores indicate severe prurigo nodularis.
Time Frame: At Weeks 2, 4, and 10
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Score on a scale
  Change from Baseline to Week 2 | -0.2 (0.52) | -0.1 (0.52)
  Change from Baseline to Week 4 | -0.4 (0.71) | -0.3 (0.71)
  Change from Baseline to Week 10 | -0.5 (0.86) | -0.4 (0.86)
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; At Week 2; Test type: Superiority; p = 0.175, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 2: Comparison: Serlopitant 5 mg vs Placebo; At Week 4; Test type: Superiority; p = 0.169, ANCOVA — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Serlopitant 5 mg vs Placebo; At Week 10; Test type: Superiority; p = 0.516, ANCOVA — [p-value comment as in outcome 4, analysis 2]

8. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) to Week 10
Description: Dermatology Life Quality Index (DLQI) is a dermatology specific quality of life (QoL) instrument designed to assess the impact of the skin disease on a subject's QoL over the prior week. It is a ten item questionnaire that assesses overall QoL and six aspects that may affect QoL (symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment). The DLQI questions are rated by the subject as 0 (not at all) to 3 (very much). Scores range from 0 to 30 with higher scores indicating poor QoL.
Time Frame: At Week 10
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Score on a scale | -4.1 (5.20) | -4.3 (5.21)
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; At Week 10; Test type: Superiority; p = 0.814, ANCOVA — [p-value comment as in outcome 4, analysis 2]

9. Secondary Outcome: Change From Baseline in DLQI Question 1 to Week 10
Description: DLQI is a dermatology specific QoL instrument designed to assess the impact of the skin disease on a subject's QoL over the prior week. It is a ten item questionnaire that assesses overall QoL and six aspects that may affect QoL (symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment) The DLQI question 1 is to measure how itchy, sore, painful or stinging the subject's skin had been. It is rated by the subject as 0 (not at all) to 3 (very much). Scores range from 0 to 30 with higher scores indicating poor QoL.
Time Frame: At Week 10
Population: Intent-to-Treat Population: included all randomized subjects who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 142 | 142
Score on a scale | -0.8 (0.80) | -0.6 (0.81)
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; At Week 10; Test type: Superiority; p = 0.113, ANCOVA — [p-value comment as in outcome 4, analysis 2]

10. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events and Serious Adverse Events (SAEs)
Description: Adverse events (AEs) and serious adverse events (SAEs) were recorded from the first study drug administration through the follow-up visit. Severity of all AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03. During the period between informed consent and first study drug dose, only SAEs caused by a protocol-mandated intervention were collected.
Time Frame: 35 days (+3 days) after Week 10 or Early Treatment Discontinuation
Population: Safety population: included all treated subjects with at least one post-baseline assessment or a reported TEAE.
Measure: Count of Participants; unit: Participants
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 139 | 141
Participants
  Subjects with any TEAE | 74 | 64
  Subjects with any Related TEAE | 20 | 9
  Subjects with any Serious TEAE | 6 | 3
  Subjects with any Related Serious TEAE | 0 | 0
  Subjects who Died | 0 | 0
  Subjects who discontinued drug due to TEAE | 5 | 3

ADVERSE EVENTS:
Time Frame: 35 days (+3 days) after Week 10 or Early Treatment Discontinuation
Description: Adverse events (AEs) and serious adverse events (SAEs) were recorded from the first study drug administration through the follow-up visit. Severity of all AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03. During the period between informed consent and first study drug dose, only SAEs caused by a protocol-mandated intervention were collected.
Arm/Group | Serlopitant 5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/141
Serious Adverse Events (participants affected / at risk) | 6/139 | 3/141
Other Adverse Events (participants affected / at risk) | 18/141 | 5/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=139) | Placebo (N=141)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=141) | Placebo (N=139)
Upper respiratory tract infection (Infections and infestations) | 10 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03546816/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03546816/SAP_001.pdf